CLINICAL TRIAL: NCT02017054
Title: Feasibility and Outcomes of Repetitive Radial Approach
Status: Withdrawn | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0827-IB-CTIL
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2016-05

CONDITIONS: Injury of Radial Artery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cath patients: Patients with previous cardiac cath via the radial access who are planned for additional radial access cardiac cath
  Interventions: Other: Cath

INTERVENTIONS:
Other: Cath — No intervention - registry
  Other Names: No intervention - registry

SUMMARY:
The purpose of this study is to assess the feasibility of performing repetitive coronary angiograms via the radial approach

DETAILED DESCRIPTION:
Assessing succes of radial access in patients with prior TRA procedures

ELIGIBILITY:
Inclusion Criteria:

Patients with previous successful radial artery approach scheduled for elective transradial coronary angiography

Exclusion Criteria:

Lack of indication to perform radial approach Abnormal Barbeau test result (type C and D) Presence of radial artery occlusion Previous important trauma of the upper limbs Presence of fistula for renal dialysis Lymphoedema Acute myocardial infarction Refusal to sign the informed consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with previous history of trans radial cardiac cath who are planned for additional trans radial cardiac cath
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To assess patency of radial artery after repetitive radial artery access | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Amit Segev, MD, Principal Investigator — Sheba MC
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel